CLINICAL TRIAL: NCT03965143
Title: Talus Replacement Registry
Acronym: 3DTalar
Status: Recruiting | Type: Observational
Sponsor: Kyle Schweser MD (Other)
Responsible Party: Sponsor-Investigator, Kyle Schweser MD, Assistant Professor Orthopaedic Trauma/Foot and Ankle, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Other Study IDs: 2014893
Record Dates: First submitted 2019-05-14; First posted 2019-05-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Avascular Necrosis of the Talus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3D talar group: Patients that will undergo a 3D custom talar augment
  Interventions: Device: 3D talar augmentation

INTERVENTIONS:
Device: 3D talar augmentation — Patients with an avascular necrosis of the body if the talar bone will undergo a 3D custom talar augmentation with or without concomitant ankle arthroplasty

SUMMARY:
Avascular necrosis of the talus is a difficult problem to manage, especially in the young and healthy. The only option, historically, has been a talectomy and hindfoot fusion. While this is a viable option, it is not without its morbidity. Arthritis of surrounding joints is common, occurring anywhere from 1-10 years after the procedure. This is especially true in younger patients, where loss of motion can be life altering both physically and mentally. The search for alternatives has been limited. Recently, 3D printing has become more ubiquitous and affordable and newer medical alternatives have arisen thanks to this technology. The 3D custom talus is relatively new in the orthopaedic community, but has been used at several centers with good success. It has been shown to re-establish the normal alignment of the foot, preserve motion (with some achieving almost physiologic motion), and allow for almost normal ambulation. However, the data is still limited and further study is necessary. Our facility was recently approved to perform this procedure. Our hypothesis is that custom 3D printed talar body replacements, either used alone or with total ankle replacements, will maintain physiologic motion, have no difference in complications when compared to hindfoot fusions with allograft, lead to good outcome scores and patient satisfaction scores. Patients diagnosed with avascular necrosis of the talus who have already decided to undergo a procedure involving a 3D custom talus as part of their standard care (talar replacement, total ankle/total talus, etc) will be enrolled in the study. Patients will follow standard post-operative protocols and return to clinic at designated time periods (2 weeks, 6 weeks, 3 months, 6 months, 1 year). X-ray evaluation, Range of motion, return to ambulation, walking speed and patient reported outcomes will be evaluated at each visit. Data will then be compared with baseline measurements and use to determine the progression of patients over time after the procedure

DETAILED DESCRIPTION:
After patients have undergone a standard of care 3D talar augment procedure they will return to clinic at designated time periods (2 weeks, 6 weeks, 3 months, 6 months, 1 year). X-rays performed as standard of care will be evaluated. Walking speed will be assessed after patient is allowed to bear weight at the same designated time periods reported above. Patients will also answer questions regarding pain (VAS survey), satisfaction (SSQ-8 survey), outcomes utilizing AAOS foot and ankle scores (survey), and self-reported return to unassisted ambulation. Goniometer measurements will be taken in the clinic at all post-operative visits to determine ROM

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 years or above at time of screening
2. Condition satisfies requirement for total talus replacement
3. Able to consent and participate in the study
4. No previous history of septic arthritis involving the hindfoot/midfoot
5. Previous ability to ambulate

Exclusion Criteria:

1. Active infection, sepsis, osteomyelitis or history of septic arthritis involving the hindfoot/midfoot
2. Unable to consent or participate in the study secondary to mental status
3. Condition does not qualify for a total talus replacement
4. Patients who are pregnant or imprisoned
5. Planned relocation or unable to return for required follow-up visits

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age diagnosed with avascular necrosis of the talar body and amenable to treatment with 3D custom augmentation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change Range of motion | 12 months
  Measures with a Goniometer and expressed in degrees
Change in VAS pain Score | 12 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Change in AAOS foot an ankle score | 12 months
  The AAOS foot and ankle questionnaire is a patient-administrated 25-item survey specifically developed for foot and ankle-related disability. The questionnaire is divided into two scales, the Foot and Ankle Core scale, comprised of 20 questions and the Shoe Comfort Scale with five questions. The questions themselves are distributed among five different categories: Pain (9 items), function (6 items), stiffness and swelling (2 items), giving way (3 items) and shoe comfort (5 items). Answers are then measured on a scale of 1 to 5 or 6, with 1 being the best outcome score.
SSQ-8 satisfaction score | 12 months
  the SSQ-8 (Surgical Satisfaction Score) is a Patient administered 8-item survey designed to asses satisfaction after a surgical procedure. Answers are then measured on a scale of 1 to 5 or 6, with 1 being the best outcome score.
Change in walking speed | 12 months
  Speed will be measured in seconds over a standard distance

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Schweser, MD, Principal Investigator — Assistant Professor Orthopaedic Trauma/Foot and Ankle
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The Investigator will maintain all study records according to applicable University regulatory requirement(s). Hard copy records will be retained for at least 7 years after the last clinic follow-up visit at the Missouri Orthopaedic Institute in a locked filing cabinet. Electronic records will be retained for the same amount of time but on secured computers and servers. If the Investigator withdraws from the responsibility of keeping the study records, custody will be transferred to a person willing to accept the responsibility.

REFERENCES:
- [Background] Jehan S, Shakeel M, Bing AJ, Hill SO. The success of tibiotalocalcaneal arthrodesis with intramedullary nailing--a systematic review of the literature. Acta Orthop Belg. 2011 Oct;77(5):644-51. PMID 22187841
- [Background] Ketz J, Myerson M, Sanders R. The salvage of complex hindfoot problems with use of a custom talar total ankle prosthesis. J Bone Joint Surg Am. 2012 Jul 3;94(13):1194-200. doi: 10.2106/JBJS.K.00421. PMID 22760387
- [Result] Wagener J, Gross CE, Schweizer C, Lang TH, Hintermann B. Custom-made total ankle arthroplasty for the salvage of major talar bone loss. Bone Joint J. 2017 Feb;99-B(2):231-236. doi: 10.1302/0301-620X.99B2.BJJ-2016-0504.R2. PMID 28148666
- [Result] Tracey J, Arora D, Gross CE, Parekh SG. Custom 3D-Printed Total Talar Prostheses Restore Normal Joint Anatomy Throughout the Hindfoot. Foot Ankle Spec. 2019 Feb;12(1):39-48. doi: 10.1177/1938640018762567. Epub 2018 Mar 14. PMID 29537314